CLINICAL TRIAL: NCT02282345
Title: A Pilot Study of Talazoparib as a Neoadjuvant Study in Patients With a Diagnosis of Invasive Breast Cancer and a Deleterious BRCA Mutation
Brief Title: Talazoparib Before Standard Therapy in Treating Patients With Invasive, BRCA-Mutated Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0045; NCI-2015-00335 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0045 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Breast Adenocarcinoma; Deleterious BRCA1 Gene Mutation; Deleterious BRCA2 Gene Mutation; HER2/Neu Negative; Invasive Breast Carcinoma
MeSH Terms: interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (talazoparib) (Experimental): Patients receive talazoparib PO QD on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then proceed to the standard of care therapy of the treating physician's choice.
  This arm was concluded early after 13 patients. An expansion arm of 20 patients was opened in August 2016 to include at least 4 and up to 6 cycles of talazoparib, followed by surgery to estimate residual cancer burden after therapy with single-agent talazoparib.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Talazoparib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673

SUMMARY:
This phase II trial studies the side effects of talazoparib when given before standard therapy in treating patients with breast cancer that has spread to nearby healthy tissue and has a mutation in a breast cancer, early onset (BRCA) gene. Talazoparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth, and may be especially effective in patients with BRCA mutations. It is not yet known whether adding talazoparib before standard treatment is safe in treating patients with BRCA mutated breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of using talazoparib prior to initiating standard neoadjuvant therapies.

II. To evaluate the toxicity profile in women taking talazoparib in the neoadjuvant setting.

SECONDARY OBJECTIVES:

I. To provide first estimate of clinical response to talazoparib in the neoadjuvant setting in a pilot trial setting.

II. To evaluate biomarkers of therapy efficacy as well as initiate patient derived xenograft (PDX) models: targeted or whole exome sequencing for BRCA pathway mutations and other somatic and germline alterations; ribonucleic acid (RNA) sequencing; evaluation of changes in immune response; transcriptional profile to assess triple negative breast cancer (TNBC) subtype, BRCA-ness signature and putative PARP sensitivity predictors; functional proteomics with reverse phase protein array (RPPA); generate PDX models and mammosphere cultures from patient derived tumors; PTEN, gamma-H2A histone family, member x (gamma-H2A.X), Ki-67 and cleaved caspase 3 by immunohistochemistry (IHC).

OUTLINE:

Patients receive talazoparib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then proceed to the standard of care therapy of the treating physician's choice.

After completion of study treatment, patients are followed up until the day after definitive breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically confirmed primary invasive adenocarcinoma of the breast with the size of the primary tumor being at least 1 cm on imaging by either mammography, ultrasound or breast magnetic resonance imaging (MRI)
* Negative human epidermal growth factor receptor 2 (HER-2)/neu- disease defined as patients with fluorescence in situ hybridization (FISH) ratio < 2.0 or < 6.0 HER2 gene copies per nucleus, and IHC staining scores of 0, 1+, or 2+
* No treatment for current primary invasive adenocarcinoma of the breast such as irradiation, chemotherapy, immunotherapy, investigational therapy or surgery; previous treatment for breast and/or ovarian cancer with chemotherapy, endocrine therapy, surgery and radiation are allowed if >= 3 years prior to current diagnosis and there is no clinical evidence of metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Baseline multi gated acquisition scan (MUGA) or echocardiogram scans with left ventricular ejection fraction (LVEF) of > 50%
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin (Hgb) >= 9 g/dL
* Creatinine clearance > 50 ml/min
* Total bilirubin =< 1.5 X upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 X ULN
* Negative serum or urine pregnancy test for women within 7 days of receiving the first dose of the study medication for women of childbearing potential; women will be considered not of childbearing potential and exempt from pregnancy testing if they are either a) older than 50 and amenorrheic for at least 12 consecutive months following cessation of all exogenous hormonal treatments, or b) have documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of investigational product; men on study also must be using contraception
* Identified deleterious mutation in BRCA 1 or 2 genes (this does not include variants of uncertain significance)
* Eligible to receive standard of care chemotherapy and/or surgery based upon standard practices or institutional guidelines

Exclusion Criteria:

* Women who are pregnant (including positive pregnancy test at enrollment or prior to study drug administration) or breast-feeding
* Disease free of prior malignancy for < 3 years with the exception of curatively treated basal carcinoma of the skin or carcinoma in situ of the cervix
* Any other previous antitumor therapies for the current cancer event
* Has had major surgery within 21 days before cycle 1 day 1
* Gastrointestinal tract disease or defect with associated malabsorption syndrome
* Uncontrolled inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* Myocardial infarction within 6 months before starting therapy, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* Serious intercurrent infections or non-malignant medical illness that are uncontrolled or the control of which may be jeopardized by this therapy
* Psychiatric disorders or other conditions rendering the subject incapable of complying with the requirements of the protocols
* Unable to take oral medications
* Known to be human immunodeficiency virus positive
* Known active hepatitis C virus, or known active hepatitis B virus
* Concurrent disease or condition that would interfere with study participation or safety, such as any of the following:

  * Active, clinically significant infection either grade > 2 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03 or requiring the use of parenteral anti-microbial agents within 14 days before day 1 of study drug
  * Clinically significant bleeding diathesis or coagulopathy, including known platelet function disorders
  * Non-healing wound, ulcer, or bone fracture
* Known hypersensitivity to any of the components of talazoparib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Litton, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kumar T, Hobbs E, Yang F, Chang JT, Contreras A, Cuentas ERP, Garber H, Lee S, Lu Y, Scoggins ME, Adrada BE, Whitman GJ, Arun BK, Mittendorf EA, Litton JK. Tumor Immune Microenvironment Changes by Multiplex Immunofluorescence Staining in a Pilot Study of Neoadjuvant Talazoparib for Early-Stage Breast Cancer Patients with a Hereditary BRCA Mutation. Clin Cancer Res. 2022 Sep 1;28(17):3669-3676. doi: 10.1158/1078-0432.CCR-21-1278. PMID 35736816
- [Derived] Litton JK, Scoggins ME, Hess KR, Adrada BE, Murthy RK, Damodaran S, DeSnyder SM, Brewster AM, Barcenas CH, Valero V, Whitman GJ, Schwartz-Gomez J, Mittendorf EA, Thompson AM, Helgason T, Ibrahim N, Piwnica-Worms H, Moulder SL, Arun BK. Neoadjuvant Talazoparib for Patients With Operable Breast Cancer With a Germline BRCA Pathogenic Variant. J Clin Oncol. 2020 Feb 10;38(5):388-394. doi: 10.1200/JCO.19.01304. Epub 2019 Aug 28. PMID 31461380
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from the breast medical oncology clinic at MD Anderson Cancer Center
Pre-assignment Details: 36 participants signed the consent, 3 participants were inevaluable
Groups:
- Talazoparib (2 Months): Talazoparib was administered as single-agent oral dose of 1 mg per day for six cycles (each cycle was 28 days) for 2 months followed by standard of care chemotherapy.
- Expansion Arm Talazoparib (6 Months) + Surgery: Talazoparib will be administered orally at 1 mg per day for at least 4 and up to 6 cycles. Each cycle will consist of 28 days (+/-3 days) followed by surgery or standard of care chemotherapy.
Period: Overall Study
Arm/Group | Talazoparib (2 Months) | Expansion Arm Talazoparib (6 Months) + Surgery
Started | 13 | 20
Completed | 13 | 19
Not Completed | 0 | 1
Not completed — Progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 patient did not go to surgery but went to chemotherapy for suspected progression
Groups:
- Talazoparib - (2 Months): Talazoparib was administered as single-agent oral dose of 1 mg per day for six cycles (each cycle was 28 days) for 2 months followed by standard of care chemotherapy.
- Expansion Arm (Talazoparib (6 Months) + Surgery): Talazoparib will be administered orally at 1 mg per day for at least 4 and up to 6 cycles. Each cycle will consist of 28 days (+/-3 days) followed by surgery or standard of care chemotherapy.
- Total: Total of all reporting groups
Arm/Group | Talazoparib - (2 Months) | Expansion Arm (Talazoparib (6 Months) + Surgery) | Total
Number analyzed (Participants) | 13 | 20 | 33
Age, Continuous [Median (Full Range); unit: years] | 40 [25 to 55] | 38 [23 to 58] | 38 [23 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 33
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 10 | 15 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 13 | 20 | 33
Number of Participants with Breast Cancer Gene and 2 (BRCA1/2) Mutations at Baseline [Count of Participants; unit: Participants]
  BRCA1 | 10 | 16 | 26
  BRCA2 | 3 | 4 | 7
Clinical stage [Count of Participants; unit: Participants] — Per the National Cancer Institute Definitions:
  Stage of Cancer.
  For Stage I, II, III, cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues
  Participants
    I | 2 | 5 | 7
    II | 9 | 12 | 21
    III | 2 | 3 | 5
Histology [Count of Participants; unit: Participants]
  Ductal | 12 | 18 | 30
  Metaplastic | 1 | 1 | 2
  Metaplastic chondrosarcomatous | 0 | 1 | 1
Chemotherapy regimen used [Count of Participants; unit: Participants]
  AC followed or preceded by weekly taxol | 13 | 0 | 13
  Addition of carboplatin to weekly taxol | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Pathological Complete Response (pCR)
Description: Pathologic response was documented using the Residual Cancer Burden (RCB) Calculator. Residual cancer burden by ICR will be reported as a categorical variable with four classes (categories) RCB 0 (pCR) which correlates to no invasive disease in breast and lymph, I (minimal RCB), II (moderate RCB), and III (extensive RCB). Up to two fine needle aspirates (FNAs) will also be obtained at each time point for a total of up to 6 FNA's for the trial, which will be used for the patient derived xenograft models. Pre-study biopsies, as well as biopsies within 7 days prior to the completion of 2 months of talazoparib will be collected via diagnostic imaging. During the expansion phase of this trial, ultrasounds will be obtained every 2 cycles (+/- 1 week). Therapy will be discontinued if the Physician or PI indicates clinically significant progression of disease.
Time Frame: Up to 6 months
Population: 1 patient did not go to surgery but went to chemotherapy for suspected progression
Measure: Count of Participants; unit: Participants
Groups:
- Talazoparib (2 Months) +(SOC) Chemotherapy: Talazoparib was administered as single-agent oral dose of 1 mg per day for six cycles (each cycle was 28 days) for 2 months followed by standard of care (SOC) chemotherapy.
Arm/Group | Talazoparib (2 Months) +(SOC) Chemotherapy | Expansion Arm Talazoparib (6 Months) + Surgery
Number analyzed (Participants) | 13 | 20
Participants
  Residual Cancer Burden 0 | 7 | 10
  Residual Cancer Burden I | 3 | 2
  Residual cancer Burden II | 3 | 5
  Residual Cancer Burden III | 0 | 2

2. Primary Outcome: Number of Participants With Grade 4 Toxicities
Description: To assess the toxicity profile of women taking single agent Talazoparib prior to surgery. If greater than 33% of the patients enrolled have either a grade 4 toxicity possibly, probably, or definitely related to the treatment as attributed by the Principal Investigator, or requires a delay in treatment for greater than 4 weeks due to toxicity.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Talazoparib - (2 Months) + (SOC) Chemotherapy.: Talazoparib was administered as single-agent oral dose of 1 mg per day for six cycles (each cycle was 28 days) for 2 months followed by standard of care (SOC)chemotherapy.
Arm/Group | Talazoparib - (2 Months) + (SOC) Chemotherapy. | Expansion Arm (Talazoparib (6 Months) + Surgery)
Number analyzed (Participants) | 13 | 20
Participants | 0 | 1

3. Secondary Outcome: Median Clinical Response to Single Agent Talazoparib
Description: Imaging was the primary measures response with tumor volume shrinkage after 2 months of Talazoparib prior to proceeding with standard chemotherapy for all participants. The clinical response to Talazoparib in the neoadjuvant setting in a pilot trial setting.
Time Frame: 2 months
Measure: Median (95% Confidence Interval); unit: percentage of tumor volume shrinkage
Groups:
- Talazoparib (2 Months): Talazoparib was administered as single-agent oral dose of 1 mg per day for six cycles (each cycle was 28 days) for 2 months followed by standard of care (SOC) chemotherapy.
Arm/Group | Talazoparib (2 Months)
Number analyzed (Participants) | 13
percentage of tumor volume shrinkage | 88 [30 to 98]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from date of consent to date patients started new treatment, an average of 1 year
Arm/Group | Talazoparib (2 Months) | Expansion Arm Talazoparib (6 Months) + Surgery
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/20
Other Adverse Events (participants affected / at risk) | 9/13 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib (2 Months) (N=13) | Expansion Arm Talazoparib (6 Months) + Surgery (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib (2 Months) (N=13) | Expansion Arm Talazoparib (6 Months) + Surgery (N=20)
Anemia (Blood and lymphatic system disorders) | 9 | 15
Leukopenia (Blood and lymphatic system disorders) | 8 | 0
Neutropenia (decreased ANC) (Blood and lymphatic system disorders) | 7 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1
Mucositis/mouth sore (Gastrointestinal disorders) | 5 | 0
Dizziness (Nervous system disorders) | 8 | 6
Fatigue (General disorders) | 7 | 14
Nausea (Gastrointestinal disorders) | 7 | 15
Elevated ALT/AST (Investigations) | 4 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
GI disorder (stomach cramps/pain) (Gastrointestinal disorders) | 3 | 0
Headache (Nervous system disorders) | 3 | 2
Hyperbilirubinemia (Blood and lymphatic system disorders) | 2 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Hypomagnesemia (Blood and lymphatic system disorders) | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 11
Constipation (Gastrointestinal disorders) | 2 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Eye redness/pain (Eye disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Blood and lymphatic system disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Decreased white blood cells (Blood and lymphatic system disorders) | 8 | 12
Neutropenia (Blood and lymphatic system disorders) | 7 | 7
Hyperglycemia (Blood and lymphatic system disorders) | 0 | 5
Pain (General disorders) | 0 | 5
Pain in breast (General disorders) | 0 | 4
Increased transaminases (General disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 0 | 3
Urinary tract infection (Renal and urinary disorders) | 0 | 3
Increased Creatinine (Investigations) | 0 | 1
Increased Phosphorous (General disorders) | 0 | 1
Increased Blood Urea Nitrogen (BUN) (Renal and urinary disorders) | 0 | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 0 | 1
Anxiety (Nervous system disorders) | 0 | 1
Vaginal Bleeding (Reproductive system and breast disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperphoshatemia (Blood and lymphatic system disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT02282345/Prot_SAP_000.pdf